CLINICAL TRIAL: NCT00925704
Title: A Phase I, Randomized, Open-Label, Three Period Cross-Over Study to Assess the Pharmacokinetics of Oral Calcitriol (ROCALTROL®) in Healthy Volunteers When Administered Alone or When Co-Administered With Lanthanum Carbonate (FOSRENOL®) or Sevelamer Carbonate (RENVELA®)
Brief Title: The Pharmacokinetics of Rocaltrol When Administered Alone or in Combination With Fosrenol or Renvela in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: SPD405-129
Record Dates: First submitted 2009-06-19; First posted 2009-06-22 (Estimated); Results first posted 2010-05-14 (Estimated); Last update posted 2021-06-15 (Actual); Status verified 2021-05

CONDITIONS: Healthy
MeSH Terms: interventions — Calcitriol; lanthanum carbonate; Sevelamer

ARMS (3):
- Calcitriol (Active Comparator)
  Interventions: Drug: Calcitriol
- Lanthanum carbonate + calcitriol (Experimental)
  Interventions: Drug: Lanthanum carbonate + Calcitriol
- Sevelamer carbonate + calcitriol (Experimental)
  Interventions: Drug: Sevelamer carbonate + Calcitriol

INTERVENTIONS:
Drug: Calcitriol — Calcitriol (1.0 microgram) single dose at lunch administered on Day 1 of the study period.
  Other Names: Rocaltrol
  Arms: Calcitriol
Drug: Lanthanum carbonate + Calcitriol — Lanthanum carbonate (1000 mg three times daily with meals for one day) + calcitriol (1.0 microgram) single dose at lunch administered on Day 1 of the study period.
  Other Names: Fosrenol + Rocaltrol
  Arms: Lanthanum carbonate + calcitriol
Drug: Sevelamer carbonate + Calcitriol — Sevelamer carbonate (2400 mg three times daily with meals for one day) + calcitriol (1.0 microgram) single dose at lunch administered on Day 1 of the study period.
  Other Names: Renvela + Rocaltrol
  Arms: Sevelamer carbonate + calcitriol

SUMMARY:
To assess the effects of lanthanum carbonate (FOSRENOL) or sevelamer carbonate (RENVELA) on the pharmacokinetics of oral calcitriol (ROCALTROL)

ELIGIBILITY:
Inclusion criteria

* Healthy volunteers age 19-45 years inclusive at the time of consent.
* Satisfactory medical assessment with no clinically significant or relevant abnormalities in medical history, physical examination, vital signs, electrocardiogram (ECG) and laboratory evaluation (hematology, biochemistry, urinalysis) as assessed by the Investigator.
* No current or recurrent disease (e.g. cardiovascular, renal, liver, gastrointestinal (GI), malignancy or other conditions) that could affect the action, absorption or disposition of the investigational products utilized in this study, or could affect clinical or laboratory assessments.

Exclusion criteria

* Current or recurrent disease (eg, cardiovascular, renal, liver, GI, malignancy or other conditions) that could affect the action, absorption or disposition of the investigational products utilized in this study, or could affect clinical or laboratory assessments.
* Current or relevant previous of physical or psychiatric illness, any medical disorder that could have required treatment or made the subject unlikely to fully complete the study, or any condition that presented undue risk from the investigational product or study procedures.
* Current use of any medication with the exception of hormonal replacement therapy or hormonal contraceptives within 14 days of first dose of investigational product.
* History of alcohol or other substance abuse within the last year.
* A positive human immunodeficiency virus antibody screen, Hepatitis B surface antigen or Hepatitis C virus antibody screen.
* Use of tobacco in any form
* Donation of blood or blood products (eg, plasma or platelets) within 60 days prior to receiving the first dose of investigational product.

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2009-06-01 (Actual); Primary Completion 2009-07-31 (Actual); Study Completion 2009-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- West Coast Clinical Trials, Cypress, California, United States

REFERENCES:
- [Result] Pierce D, Hossack S, Poole L, Robinson A, Van Heusen H, Martin P, Smyth M. The effect of sevelamer carbonate and lanthanum carbonate on the pharmacokinetics of oral calcitriol. Nephrol Dial Transplant. 2011 May;26(5):1615-21. doi: 10.1093/ndt/gfq598. Epub 2010 Oct 4. PMID 20921291
- See also: FDA recall information — http://www.fda.gov/opacom/7alerts.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients were randomly assigned to 1 of 6 treatment sequences which consisted of 3 treatment periods separated by a washout of 7 days. In each of the treatment periods subjects received lanthanum carbonate + calcitriol, sevelamer carbonate + calcitriol or calcitriol alone.
Groups:
- Sequence 1: Calcitriol (1.0 microgram) single dose at lunch for one day in first intervention, washout, Lanthanum carbonate (1000 mg three times daily with meals) + Calcitriol (1 microgram single dose at lunch) for one day in second intervention, washout, Sevelamer carbonate (2400 mg three times daily with meals) + Calcitriol (1 microgram single dose at lunch) for one day in third intervention
- Sequence 2: Lanthanum carbonate (1000 mg three times daily with meals) + Calcitriol (1 microgram single dose at lunch) for one day in first intervention, washout, Calcitriol (1.0 microgram) single dose at lunch for one day in second intervention, washout, Sevelamer carbonate (2400 mg three times daily with meals) + Calcitriol (1 microgram single dose at lunch) for one day in third intervention
- Sequence 3: Lanthanum carbonate (1000 mg three times daily with meals) + Calcitriol (1 microgram single dose at lunch) for one day in first intervention, washout, Sevelamer carbonate (2400 mg three times daily with meals) + Calcitriol (1 microgram single dose at lunch) for one day in second intervention, washout, Calcitriol (1.0 microgram) single dose at lunch for one day in third intervention
- Sequence 4: Sevelamer carbonate (2400 mg three times daily with meals) + Calcitriol (1 microgram single dose at lunch) for one day in first intervention, washout, Calcitriol (1.0 microgram) single dose at lunch for one day in second intervention, washout, Lanthanum carbonate (1000 mg three times daily with meals) + Calcitriol (1 microgram single dose at lunch)for one day in third intervention
- Sequence 5: Sevelamer carbonate (2400 mg three times daily with meals) + Calcitriol (1 microgram single dose at lunch) for one day in first intervention, washout, Lanthanum carbonate (1000 mg three times daily with meals) + Calcitriol (1 microgram single dose at lunch) for one day in second intervention, washout, Calcitriol (1.0 microgram) single dose at lunch for one day in third intervention
- Sequence 6: Calcitriol (1.0 microgram) single dose at lunch for one day in first intervention, washout, Sevelamer carbonate (2400 mg three times daily with meals) + Calcitriol (1 microgram single dose at lunch) for one day in second intervention, washout, Lanthanum carbonate (1000 mg three times daily with meals) + Calcitriol (1 microgram single dose at lunch)for one day in third intervention
Period: First Intervention
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 6 | 7 | 7 | 7 | 7 | 7
Completed | 6 | 7 | 7 | 6 | 6 | 7
Not Completed | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Withdrew consent | 0 | 0 | 0 | 1 | 1 | 0
Period: Washout
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 6 | 7 | 7 | 6 | 6 | 7
Completed | 6 | 7 | 7 | 6 | 6 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 6 | 7 | 7 | 6 | 6 | 7
Completed | 5 | 7 | 7 | 6 | 5 | 7
Not Completed | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 1 | 0
Period: Washout
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 5 | 7 | 7 | 6 | 5 | 7
Completed | 5 | 7 | 7 | 6 | 5 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 5 | 7 | 7 | 6 | 5 | 7
Completed | 5 | 7 | 7 | 6 | 5 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrew consent | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Total
Number analyzed (Participants) | 6 | 7 | 7 | 7 | 7 | 7 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 7 | 7 | 7 | 7 | 7 | 41
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.7 (8.94) | 30.0 (6.24) | 30.9 (5.52) | 28.4 (7.28) | 31.0 (8.52) | 30.4 (10.41) | 29.8 (7.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 2 | 2 | 4 | 3 | 19
  Male | 1 | 4 | 5 | 5 | 3 | 4 | 22
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 7 | 7 | 7 | 7 | 7 | 41

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Serum Concentration-time Curve (AUC 0-48) for Exogenous Calcitriol
Description: This shows the effect that lanthanum carbonate or sevelamer carbonate has on the pharmacokinetics of oral calcitriol. Exogenous calcitriol was the difference between total calcitriol value and the baseline exogenous calcitriol value at each sampling timepoint.
Time Frame: pre-dose, 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36, and 48 hours post calcitriol dose
Population: Pharmacokinetic set (PK) consists of subjects who received at least 1 dose of investigational product, had evaluable serum concentration-time profiles for calcitriol through 48 hours post-dosing on Day 1 of any treatment period and did not vomit between dosing and 10 hours post-dose on Day 1 of that treatment period.
Measure: Least Squares Mean (95% Confidence Interval); unit: pg*h/ml
Groups:
- Calcitriol (Lanthanum Carbonate): This group is the least squares mean of AUC 0-48 Lanthanum carbonate + Calcitriol minus least squares mean of AUC 0-48 Calcitriol alone.
- Calcitriol (Sevelamer Carbonate): This group is the least squares mean of AUC 0-48 Sevelamer carbonate + Calcitriol minus least squares mean of AUC 0-48 Calcitriol alone.
Arm/Group | Calcitriol (Lanthanum Carbonate) | Calcitriol (Sevelamer Carbonate)
Number analyzed (Participants) | 41 | 41
pg*h/ml | 111 [-48.9 to 270] | -181 [-338 to -24.0]
Statistical Analysis 1: Comparison: Calcitriol (Lanthanum Carbonate); Exogenous calcitriol was analyzed using a mixed linear effects model. This model contained sequence group, period, and treatment as fixed effects. The subject within sequence effect was included as a random effect; Test type: Superiority or Other; p = 0.171, Mixed Models Analysis
Statistical Analysis 2: Comparison: Calcitriol (Sevelamer Carbonate); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.024, Mixed Models Analysis

2. Secondary Outcome: Maximum Plasma Concentration (Cmax) for Exogenous Calcitriol
Description: as for outcome 1
Time Frame: pre-dose, 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36, and 48 hours post calcitriol dose
Population: PK set
Measure: Least Squares Mean (95% Confidence Interval); unit: pg/ml
Groups:
- Calcitriol (Lanthanum Carbonate): This group is the least squares mean of Cmax Lanthanum carbonate + Calcitriol minus least squares mean of Cmax Calcitriol alone.
- Calcitriol (Sevelamer Carbonate): This group is the least squares mean of Cmax Sevelamer carbonate + Calcitriol minus least squares mean of Cmax Calcitriol alone.
Arm/Group | Calcitriol (Lanthanum Carbonate) | Calcitriol (Sevelamer Carbonate)
Number analyzed (Participants) | 41 | 41
pg/ml | -2.74 [-8.12 to 2.63] | -9.62 [-14.9 to -4.34]
Statistical Analysis 1: Comparison: Calcitriol (Lanthanum Carbonate); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.313, Mixed Models Analysis
Statistical Analysis 2: Comparison: Calcitriol (Sevelamer Carbonate); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis

3. Secondary Outcome: Time of Maximum Plasma Concentration (Tmax) for Exogenous Calcitriol
Description: as for outcome 1
Time Frame: pre-dose, 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36, and 48 hours post calcitriol dose
Population: PK set
Measure: Median (95% Confidence Interval); unit: hours
Groups:
- Calcitriol (Lanthanum Carbonate): This group is the median of Tmax Lanthanum carbonate + Calcitriol minus the median of Tmax Calcitriol alone.
- Calcitriol (Sevelamer Carbonate): This group is the median of Tmax Sevelamer carbonate + Calcitriol minus the median of Tmax Calcitriol alone.
Arm/Group | Calcitriol (Lanthanum Carbonate) | Calcitriol (Sevelamer Carbonate)
Number analyzed (Participants) | 41 | 41
hours | 1.27 [0.00 to 2.48] | 0.500 [0.00 to 1.46]
Statistical Analysis 1: Comparison: Calcitriol (Lanthanum Carbonate); Analysis for Tmax used the Hodges-Lehmann estimate for Wilcoxon's Signed Rank Test; Test type: Superiority or Other; p = 0.039, Wilcoxon (Hodges-Lehmann)
Statistical Analysis 2: Comparison: Calcitriol (Sevelamer Carbonate); Analysis for Tmax used the Hodges-Lehmann estimate for Wilcoxon's Signed Rank Test; Test type: Superiority or Other; p = 0.305, Wilcoxon (Hodges-Lehmann)

ADVERSE EVENTS:
Description: Safety Set consisted of all enrolled subjects who received at least 1 dose of investigational product and had at least 1 post-dose safety assessment.
Groups:
- Lanthanum Carbonate + Calcitriol: Lanthanum carbonate (1000 mg three times daily with meals for one day) + Calcitriol (1 microgram single dose at lunch)
- Sevelamer Carbonate + Calcitriol: Sevelamer carbonate (2400 mg three times daily with meals for one day) + Calcitriol (1 microgram single dose at lunch)
- Calcitriol Alone: Calcitriol (1.0 microgram) single dose at lunch
Arm/Group | Lanthanum Carbonate + Calcitriol | Sevelamer Carbonate + Calcitriol | Calcitriol Alone
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/40 | 0/38
Other Adverse Events (participants affected / at risk) | 5/38 | 2/40 | 3/38
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lanthanum Carbonate + Calcitriol (N=38) | Sevelamer Carbonate + Calcitriol (N=40) | Calcitriol Alone (N=38)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 | 0
Headache (Nervous system disorders) | 2 (2) | 2 (2) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.